CLINICAL TRIAL: NCT02022644
Title: A Phase I Study of Convection-Enhanced Delivery of Liposomal-Irinotecan Using Real-Time Imaging With Gadolinium In Patients With Recurrent High Grade Glioma
Brief Title: Study of Convection-Enhanced, Image-Assisted Delivery of Liposomal-Irinotecan In Recurrent High Grade Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Ipsen (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Nicholas Butowski, Assistant Professor of Neurological Surgery; Director of Clinical Services, Division of Neuro-Oncology, University of California, San Francisco
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Nano CED; 13-12025 (Other: University of California, San Francisco); 5R21CA186140-02 (NIH); NCI-2017-01304 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP)); 13108 (Other: University of California, San Francisco)
Record Dates: First submitted 2013-12-11; First posted 2013-12-30 (Estimated); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: High Grade Glioma
MeSH Terms: conditions — Glioma | interventions — irinotecan sucrosofate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Group 1 - 20 mg (Experimental): Tumor diameter: 1 cm, Tumor volume: ~0.5cm3, Infusion Volume: 2-3 ml, Irinotecan conc.: 20 mg/ml, Infusion time: 6-24 hours, no more than 48
  Interventions: Drug: nanoliposomal irinotecan
- Group 2 - 40 mg (Experimental): Tumor diameter: 2 cm,Tumor volume: ~4.1cm3, Infusion Volume: 3-4 ml, Irinotecan conc.: 40 mg/ml, Infusion Time: 6-24 hours, no more than 48
  Interventions: Drug: nanoliposomal irinotecan
- Group 3 - 140 mg (Experimental): Tumor diameter: 3 cm, Tumor volume: ~14cm3, Infusion Volume: 6-7 ml, Irinotecan conc.: 140 mg/ml, Infusion Time: 6-24 hours, no more than 48
  Interventions: Drug: nanoliposomal irinotecan
- Group 4 - 340 mg (Experimental): Tumor diameter: 4 cm, Tumor volume: ~34cm3, Infusion Volume: ≤17 ml, Irinotecan conc.: 340 mg/ml, Infusion Time: 6-24 hours, no more than 48
  Interventions: Drug: nanoliposomal irinotecan
- Group 5 - 40 mg (Experimental): Tumor diameter: 1 cm, Tumor volume: ~0.5cm3, Infusion Volume: 2-3 ml, Irinotecan conc.: 40 mg/ml, Infusion Time: 6-24 hours, no more than 48
  Interventions: Drug: nanoliposomal irinotecan
- Group 6 - 80 mg (Experimental): Tumor diameter: 2 cm, Tumor volume: ~4.1cm3, Infusion Volume: 3-4 ml, Irinotecan conc.: 80 mg/ml, Infusion Time: 6-24 hours, no more than 48
  Interventions: Drug: nanoliposomal irinotecan
- Group 7 - 280 mg (Experimental): Tumor diameter: 3 cm, Tumor volume: ~14cm3, Infusion Volume: 6-7 ml, Irinotecan conc.: 280 mg/ml, Infusion Time: 6-24 hours, no more than 48
  Interventions: Drug: nanoliposomal irinotecan
- Group 8 - 680 mg (Experimental): Tumor diameter: 4 cm, Tumor volume: ~34cm3, Infusion Volume: ≤17 ml, Irinotecan conc.: 680 mg/ml, Infusion Time: 6-24 hours, no more than 48
  Interventions: Drug: nanoliposomal irinotecan

INTERVENTIONS:
Drug: nanoliposomal irinotecan — The drug named here (nanoliposomal irinotecan) will be used in varying amounts, based on tumor volume.
  Other Names: MM-398; ONIVYDE

SUMMARY:
This is a single center, dose-toleration study designed to investigate and determine the maximum tolerated dose of nanoliposomal irinotecan in adults with recurrent high-grade glioma when administered directly into the tumor using a process called convection-enhanced delivery (CED).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety and tolerability of liposomal-irinotecan with gadolinium given by intra tumoral real-time convection enhanced delivery in patients with recurrent high grade glioma (HGG).

SECONDARY OBJECTIVES:

I. To optimize the magnetic resonance image-guided intracranial injection procedure in patients with recurrent HGG by correlating the observed distribution of gadolinium to pre-treatment modeling of the drug distribution utilizing predictive imaging software.

EXPLORATORY OBJECTIVES:

I. To estimate the time to progression and overall survival measured from the date of CED.

II. To determine the objective tumor response rate, based upon MR imaging, every 8 weeks for first year and then every 12 weeks.

III. To evaluate the possible effect on tumor histology, as assessed by comparing pre-treatment tumor samples to post-treatment tumor samples in patients who undergo subsequent repeat surgical procedures for progression after being treated as part of this protocol.

IV. Pharmacokinetics measurements will also be taken at pre-dose, 1 day after the drug is administered, and 1 week post-op.

OUTLINE:

Participants will be enrolled in a 3+3 dose escalation model with a two cohort concentration escalation, enrolling at least 3 patients in each cohort which results in each total dose personalized for each participant as all participants will have different size and morphology of tumors requiring different volumes of study infusions ranging from 3 mL for smallest tumor to approximately 17 mL for largest tumor (4 cm). Enrollment into a subsequent cohort will not start until after 30 days after monitoring all patients in cohort prior. Participants will be followed for 12 months from CED procedure or until death or institution of alternate anti-neoplastic therapy for progressive recurrent HGG.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with radiographically proven recurrent, intracranial high grade glioma will be eligible for this protocol. Patients must have evidence of tumor progression as determined by the Revised Assessment in Neuro-Oncology RANO criteria following standard therapy.

   1. High grade glioma includes glioblastoma multiforme (GBM), Gliosarcoma (GS), anaplastic astrocytoma (AA), anaplastic oligodendroglioma (AO), anaplastic mixed oligoastrocytoma (AMO), or malignant astrocytoma not otherwise specified. (NOS)
   2. Magnetic resonance imaging (MRI) must be performed within 21 days prior to enrollment, and patients who are receiving steroids must be stable or decreasing for at least 5 days prior to imaging. If the steroid dose is increased between the date of imaging and enrollment, a new baseline MRI is required.
   3. Patients must have completed only 1 prior course of radiation therapy and must have experienced an interval of greater than 12 weeks from the completion of radiation therapy to study entry.
2. Patients will be eligible if the original histology was low-grade glioma and a subsequent histological diagnosis of a high grade glioma is made.
3. There is no limit as to the number of prior treatments but patients must have radiographic evidence of progressive disease
4. Recurrent tumor must be a solid, single, supratentorial, contrast-enhancing HGG which have a tumor diameter no larger than 4cm or volume of 34cm3
5. All patients must sign an informed consent indicating that they are aware of the investigational nature of this study.

   a. Patients must be> 18 years old, and with a life expectancy > 8 weeks
6. Patients with Karnofsky performance status of >= 70.
7. At the time of registration: Patients must have recovered from the toxic effects of prior therapy: > 10 days from any noncytotoxic investigational agent, >28 days from prior cytotoxic therapy or Avastin, >14 days from vincristine, >42 days from nitrosoureas, >21 days from procarbazine administration, and >7 days for non-cytotoxic agents, e.g., interferon, tamoxifen, thalidomide, cis-retinoic acid, etc. (radiosensitizer does not count). Any questions related to the definition of non-cytotoxic agents should be directed to the Study Chair.
8. Requirements for organ and marrow function as follows:

   1. Adequate bone marrow function:

      * leukocytes > 3,000/microliter (mcL)
      * absolute neutrophil count > 1,500/mcL
      * platelets > 100,000/mcL
   2. Adequate hepatic function:

      * total bilirubin within normal institutional limits
      * aspartate aminotransferase (AST) < 2.5 X institutional upper limit of normal
      * alanine aminotransferase (ALT) < 2.5 X institutional upper limit of normal
   3. Adequate renal function:

      * creatinine within normal institutional limits OR
      * creatinine clearance > 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal.
   4. Adequate coagulation function

      * International Normalized Ratio (INR) < 2.0
      * partial thromboplastin time (PTT) <= institution's upper limit of normal, unless receiving therapeutic low molecular weight heparin.
9. The effects of nano liposomal irinotecan on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception: hormonal or barrier method of birth control; abstinence, etc. prior to study entry, for the duration of study participation, and for 6 months post drug administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
10. Women of childbearing potential must have a negative beta-human chorionic gonadotropin (beta-HCG) pregnancy test documented within 14 days prior to treatment.
11. Patients with prior therapy that included interstitial brachytherapy, or Gliadel wafers must have confirmation of true progressive disease rather than radiation necrosis based upon either Positron Emission Tomography (PET) or Thallium scanning, MR spectroscopy or surgical documentation of disease
12. Patients must be able to have MRI brain imaging.
13. UGT1A1 genotyping will be sent for testing at screening, but results do not have to be known before starting treatment

Exclusion Criteria:

1. Patients must not have any significant medical illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy
2. Patients with a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission and off of all therapy for that disease for a minimum of 3 years are ineligible.
3. HIV-positive patients on combination antiretroviral therapy are ineligible.
4. Contrast-enhancing tumor which crosses the midline.
5. Multi-focal disease.
6. Nonparenchymal tumor dissemination (e.g., subependymal or leptomeningeal)
7. History of hypersensitivity reactions to products containing irinotecan (irinotecan), topotecan or other topoisomerase inhibitors, gadolinium contrast agents or lipid products.
8. Ongoing treatment with cytotoxic therapy.
9. Patients may not be on an enzyme-inducing anti-epileptic drug (EIAED). If previously on an EIAED, patient must be off for at least 10 days prior to CED infusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-10-23 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 30 days post-infusion
  Dose limiting toxicity (DLT) will be defined as any grade-3 or higher neurological toxicity felt to be attributable to the CED infusion of liposomal-irinotecan with gadolinium, as well as any systemic grade-3 or higher hematologic or non-hematologic toxicity (after maximal medical management of nausea/vomiting/diarrhea), over a period of 30 days after CED infusion.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) at 6 months | Up to 6 months
  Number of patients not having objective progression or death at 6 months after the time from date of study enrollment estimated from the PFS distribution. For patients who are not known to have died or progressed as of the data-inclusion cut-off date, PFS time will be censored at the date of the last objective progression-free disease assessment prior to the date of any subsequent systematic anticancer therapy. PFS will be summarized using Kaplan Meier methods and displayed graphically. The median event time and two-sided 95% confidence interval for the median will be reported.
Progression-Free Survival (PFS) | Up to 10 years
  The time from the date of study enrollment to the date of first observation of objective progression or death from any cause, whichever occurs first. For patients who are not known to have died or progressed as of the data-inclusion cut-off date, PFS time will be censored at the date of the last objective progression-free disease assessment prior to the date of any subsequent systematic anticancer therapy. PFS will be summarized using Kaplan Meier methods and displayed graphically. The median event time and two-sided 95% confidence interval for the median will be reported.
Overall Survival at 12 months | Up to 12 months
  The time from the date of study enrollment to the date of death from any cause. For patients who are not known to have died as of the 12 month cut-off date, survival time will be censored at the date of the last known survival status of participant prior to the date of any subsequent systematic anticancer therapy. OS will be summarized using Kaplan Meier methods and displayed graphically. The median event time and two-sided 95% confidence interval for the median will be reported.
Overall Survival (OS) | Up to 10 years
  The time from the date of study enrollment to the date of death from any cause. For patients who are not known to have died as of the data-inclusion cut-off date, survival time will be censored at the date of the last known survival status of participant prior to the date of any subsequent systematic anticancer therapy. OS will be summarized using Kaplan Meier methods and displayed graphically. The median event time and two-sided 95% confidence interval for the median will be reported.
Objective Tumor Response Rate | Up to 10 years
  Overall response rate (ORR) is the proportion of patients who achieved a complete response (CR) or partial response (PR) out of all randomly assigned patients. Based on Response assessment in neuro-oncology criteria (RANO), a responder is defined by radiographic and clinical criteria. Complete response or PR will be first assessed by radiographic changes as determined by an improvement of the bi-dimensional evaluation of the tumor size. In addition, changes in neurologic function and steroid use will be considered to determine stable disease (SD). The objective response rate (ORR) will be summarized with the corresponding exact two-sided 95% confidence interval calculated using a method based on the F distribution

OTHER OUTCOMES:
Pre-infusion modeling of the drug distribution vs. post-infusion imaging. | Up to 48 hours pre-infusion and up to 48 hours post-infusion
  Pre-operative MRIs will be compared to post-operative MRIs to determine the location and pattern of infusate spread.
Ratio of the Volume of distribution (Vd) to volume infused (Vi) | Up to 24 hours from time of dosing
  The volume of distribution of study infusion will be compared to the total volume infused. An average Vd/Vi will be established for each flow rate, and mean distribution volume lengths, widths, and positions with respect to the infusion cannula tip will be generated as a function of infusion volume (Vi)
Change in Tumor Histology | Up to 12 months from date of surgery
  Assessed by comparing pre-treatment tumor samples to post-treatment tumor samples in patients who undergo subsequent repeat surgical procedures. (If applicable)
Mean plasma levels of total Liposomal-irinotecan (MM-398, ONIVYDE) | Pre-infusion, 1 hour post-infusion, and approximately 1 week post-infusion
  Pharmacokinetic testing will be performed on plasma levels of total Liposomal-irinotecan (MM-398, ONIVYDE) will be measured at 0 (pre-infusion), approximately 1-hour after infusion, and approximately 1-week following the end of irinotecan infusion into the brain.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Butowski, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2020-09-28): https://cdn.clinicaltrials.gov/large-docs/44/NCT02022644/ICF_000.pdf